CLINICAL TRIAL: NCT05122689
Title: Influence of Exogenous Dietary Inorganic Nitrate on Downstream Metabolites of the Enteral Microbiome
Brief Title: Dietary Inorganic Nitrate and the Enteral Microbiome
Acronym: DINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Dietary nitrate and microbiome
Record Dates: First submitted 2021-09-10; First posted 2021-11-17 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Health
Keywords: microbiome; nitrate; diet; dietary nitrate; cardiovascular
MeSH Terms: interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate (Experimental): Dietary inorganic nitrate (0,12 mmol sodium-nitrate/kg BW/day) dissolved in 200 ml tap water. Supplementation for 30 days.
  Interventions: Dietary Supplement: Nitrate
- Control (Placebo Comparator): Dietary sodium-chloride (0,12 mmol sodium-chloride/kg BW/day) dissolved in 200 ml tap water. Supplementation for 30 days.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Nitrate — Dietary inorganic nitrate (0,12 mmol sodium-nitrate/kg BW/day) dissolved in 200 ml tap water. Supplementation for 30 days.
  Arms: Nitrate
Dietary Supplement: Control — Dietary sodium-chloride (0,12 mmol sodium-chloride/kg BW/day) dissolved in 200 ml tap water. Supplementation for 30 days.
  Arms: Control

SUMMARY:
A growing body of data shows that the enteral microbiome has an effect on cardiovascular diseases. Exogenous inorganic dietary nitrate mediates cardioprotective effects and has been shown to have an influence on the oral microbiome. The nutritional aspects of these cardioprotective effects are particularly intriguing since nitrate is abundant in our everyday diet.

Whether dietary nitrate influences the enteral microbiome and downstream metabolites like short-chain fatty acids (SCFA) and TMAO will be investigated in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 years
* no regular medication intake
* no chronic diseases

Exclusion Criteria:

* Regular systemic drug intake
* Active smoking
* Chronic diseases
* Acute diarrhea or vomiting
* Short gut syndrome
* Pregnancy or breastfeeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change of the enteral microbiome composition | 30 days
  Changes in enteral microbiome composition in stool samples at baseline and after 30 days of placebo/verum supplementation. The 16S rRNA amplicon reads obtained from an Illumina MiSeq System will be analyzed using pipeline QIIME2 (v. 2019.1).

SECONDARY OUTCOMES:
Change of the oral microbiome composition | 30 days
  Changes in oral microbiome composition in oral swabs samples at baseline and after 30 days of placebo/verum supplementation. The 16S rRNA amplicon reads obtained from an Illumina MiSeq System will be analyzed using pipeline QIIME2 (v. 2019.1).
Change of circulating SCFA levels | 30 days
  Changes in circulating SCFA blood levels at baseline and after 30 days of placebo/verum supplementation will be measured by high-performance liquid chromatography.

OTHER OUTCOMES:
Changes in the oral-enteral microbiome axis | 30 days
  Changes in oral-enteral microbiome axis composition in oral swabs and stool samples at baseline and after 30 days of placebo/verum supplementation. The 16S rRNA amplicon reads obtained from an Illumina MiSeq System will be analyzed using pipeline QIIME2 (v. 2019.1).
Changes in arterial stiffness parameters | 30 days
  Changes in cardiovascular function measured by arterial stiffness parameters as pulse wave velocity measured in m/s at baseline and after 30 days of placebo/verum supplementation.
Changes in blood pressure | 30 days
  Changes in cardiovascular function measured by systolic and diastolic blood pressure in mmHg at baseline and after 30 days of placebo/verum supplementation.
Change of the nitrate-nitrite-NO metabolism | 30 days
  Changes of nitrate and nitrite content in plasma measured by ENO-20 analysis at baseline and after 30 days of placebo/verum supplementation.
Genetic variants (single nucleotide polymorphism) | 30 days
  The effect of the genes NOS3 and GUCY1A3 variation on dietary nitrate response. Genetic polymorphism will be measured by qPCR and analyzed by allelic discrimination.
Epigenetic changes | 30 days
  Changes of DNA methylation analysis by pyrosequencing at baseline and after 30 days of placebo/verum supplementation.
Changes in TMAO levels | 30 days
  Changes in TMAO blood levels at baseline and after 30 days of placebo/verum supplementation will be measured by ultra-high-performance liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, Professor, Study Director — Clinic of cardiology and angiology, University Hospital Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Messiha D, Lange E, Tratnik A, M Westendorf A, Rinke M, Lenz S, Hendgen-Cotta UB, Buer J, Rassaf T, Rammos C. The influence of acute and chronic coronary syndrome on the gut microbiome and downstream microbiome-derived metabolites-Microbiome in acute myocardial infarction-MIAMI-Trial. Basic Res Cardiol. 2025 Oct;120(5):913-924. doi: 10.1007/s00395-025-01134-9. Epub 2025 Aug 13. PMID 40804540